CLINICAL TRIAL: NCT03260426
Title: Prospective Randomized Controlled Trial Investigating Commencement of Low Residue Diet Versus Clear Liquids on Postoperative Zero Following Elective Colorectal Surgery
Brief Title: Trial of Low Residue Diet Versus Clear Liquids Following Elective Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Clinical Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048403
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Nausea/Vomiting
Keywords: Tolerability diet after surgery
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Clear Liquid Diet (Experimental): Clear liquids on postoperative day zero and intestinal rate measured by Abstats
  Interventions: Dietary Supplement: Clear Liquids; Device: Abstats
- Regular Solid Diet (Experimental): Regular diet from postoperative day zero and intestinal rate measured by Abstats
  Interventions: Dietary Supplement: Regular Solid; Device: Abstats

INTERVENTIONS:
Dietary Supplement: Clear Liquids — Clear liquids on postoperative day zero immediately upon return to the floor and subsequent days' advancement of enteral diet to regular diet is as per discretion of the attending physician.
  Arms: Clear Liquid Diet
Dietary Supplement: Regular Solid — Regular diet from postoperative day zero immediately upon return to floor and onwards
  Arms: Regular Solid Diet
Device: Abstats — Intestinal rate measured by Abstats™ in patients offered immediate solid versus clear liquids after colorectal surgery

SUMMARY:
Prospective randomized controlled trial investigating commencement of low residue diet versus clear liquids on postoperative zero following elective colorectal surgery, with regards to patient tolerability, incidence of nausea and/or vomiting, and postoperative length of hospitalization stay.

DETAILED DESCRIPTION:
Offering patients, a low residue diet on the first postoperative day (POD1) after colorectal surgery is safe and improves surgical outcomes and postoperative hospital stay. Early use of low solid is superior to clear liquid diet after elective colorectal surgery.

The purpose of this study is to prospectively evaluate whether providing a patient a solid diet from postoperative day zero is superior to clear liquids. The primary endpoint measured will be patient tolerability, as evidenced by absence of vomiting. The secondary endpoints measured will be duration of supplemental intravenous hydration needed, length of hospital stay and postoperative complications, and intestinal rate measured by Abstats.

Abstats™ consists of a disposable plastic device embedded with a microphone that adheres to the abdominal wall and connects to a computer measuring acoustic event rates. The monitor will be placed on the patient's abdomen 30 minutes prior to surgery in the preoperative holding area to obtain baseline intestinal rate. The monitor will be removed prior to surgery and replaced by the surgical team in the operating room and maintained until postoperative day 3. Daily intestinal rate will be calculated as mean and median acoustic events per minute. The raw data will be analyzed by an investigator blinded to the clinical data. Intestinal rates of patients offered immediate solid feeds will be compared with those offered clear feeds. In addition, patients not tolerating or consuming early solid meal will be compared with those who do to identify whether Abstat™ can be an early predictor of diet intolerance in patients undergoing colorectal surgery.

Patients will be assigned into one of two groups:

Group I - Clear liquids on postoperative day zero immediately upon return to the floor and subsequent days' advancement of enteral diet to regular diet is as per discretion of the attending physician.

Group II - Regular diet from postoperative day zero immediately upon return to floor and onwards.

Three questionnaires assessing quality of life are to be completed by the patient, during his/her hospital stay. On postoperative day one, a self-administered questionnaire is to be completed by the patient. Please see appendix A for the questionnaire details. The same questionnaire is administered on postoperative day two and again on the last day of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
2. Males or females, >18 years of age inclusive at the time of study screening;
3. American Society of Anesthesiologists (ASA) Class I-III;
4. Colorectal surgery (open and/or robotic/laparoscopic);
5. Elective Surgery

Exclusion Criteria:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures.
2. Children <18 years of age.
3. Pre-operative clinical diagnosis of intestinal obstruction.
4. Pre-existing known upper gastrointestinal disorders including hiatus hernia, gastroesophageal reflux disease, peptic ulcer disease.
5. Pre-existing oropharyngeal disorders such as stomatitis, altered taste sensations.
6. Colorectal surgery with concomitant resectional surgery of the stomach or proximal jejunum (small bowel).
7. Pregnant patients.
8. Bedbound or moribund patients.
9. Pre-existing history of clinical depression.
10. Epidural analgesia.
11. Surgical procedures completed after 4pm
12. Patients taking narcotics prior to elective colorectal surgery

Exclusion Criteria After randomization:

1. Postoperative diagnosis of intra-abdominal sepsis, including anastomotic leaks.
2. Postoperative complications requiring early reoperation within the same hospital stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Fleshner, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Lau C, Phillips E, Bresee C, Fleshner P. Early use of low residue diet is superior to clear liquid diet after elective colorectal surgery: a randomized controlled trial. Ann Surg. 2014 Oct;260(4):641-7; discussion 647-9. doi: 10.1097/SLA.0000000000000929. PMID 25203881
- [Background] Spiegel BM, Kaneshiro M, Russell MM, Lin A, Patel A, Tashjian VC, Zegarski V, Singh D, Cohen SE, Reid MW, Whitman CB, Talley J, Martinez BM, Kaiser W. Validation of an acoustic gastrointestinal surveillance biosensor for postoperative ileus. J Gastrointest Surg. 2014 Oct;18(10):1795-803. doi: 10.1007/s11605-014-2597-y. Epub 2014 Aug 5. PMID 25091837
- [Derived] Yao LY, Gough AE, Zaghiyan KN, Fleshner PR. Prospective Randomized Trial of Immediate Postoperative Use of Regular Diet Versus Clear Liquid Diet in Major Colorectal Surgery. Dis Colon Rectum. 2023 Dec 1;66(12):1547-1554. doi: 10.1097/DCR.0000000000002737. Epub 2023 Aug 31. PMID 37656683

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clear Liquid Diet | Regular Solid Diet | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (50) | 45.5 (50) | 46.5 (100)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 50 | 50 | 100
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (4.3) | 22.7 (4.9) | 23.1 (4.1)
Prior abdominal surgery [Count of Participants; unit: Participants] | 21 | 20 | 41
Site of surgery [Count of Participants; unit: Participants]
  Small bowel | 9 | 12 | 21
  Right colon | 13 | 12 | 25
  Subtotal/left | 14 | 9 | 23
  pelvis | 14 | 17 | 31
Diagnosis [Count of Participants; unit: Participants]
  IBD | 39 | 37 | 76
  Cancer | 8 | 6 | 14
  Other | 3 | 7 | 10
Ostomy Use [Count of Participants; unit: Participants] — Population: Out of the 100 patients total of 49 patients received an ostomy. at the time of surgery.
  46 patient received and ileostomy and 3 patients received a colostomy.
  Participants
    Ileostomy | 24 | 22 | 46
    Colostomy | 2 | 1 | 3
    No ostomy | 24 | 27 | 51
Anastomosis [Count of Participants; unit: Participants] — Out of the 100 patients who were enrolled and had surgery only 71 patients had an anastomosis formed. That is why the total is 71 patient. 35 in clear liquid group and 36 in regular diet group had an anastomosis formed.
  Participants
    Anastomosis formed | 35 | 36 | 71
    No Anastomosis | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Emesis on Post Operative Day 2
Description: Patient tolerability, as evidenced by development of vomiting on postoperative day two.
Time Frame: POD 2
Population: All participants undergoing surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
Participants | 9 | 9

2. Secondary Outcome: Number of Participants Able to Tolerate a Regular Diet as Compared to a Clear Liquid Diet on Post Operative Day 0 (POD 0).
Description: Tolerability of regular diet will be determined by the patients ability to eat more than 50% of a solid meal on post operative day zero.
Time Frame: POD 0
Population: All participants undergoing surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
Participants | 46 | 34

3. Secondary Outcome: Antiemetic Usage
Description: If antiemetics were used in
Time Frame: 30 days
Population: All participants undergoing surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
Participants | 37 | 30

4. Secondary Outcome: Hospital Stay
Description: Length of postoperative stay
Time Frame: 30 days
Measure: Mean (Standard Error); unit: days
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
days | 3 (3.5) | 2.5 (4.0)

5. Secondary Outcome: Post-operative Ileus
Description: Development of post-operative ileus
Time Frame: 30 days
Population: All participants undergoing surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
Participants | 11 | 11

6. Secondary Outcome: Pain Score
Description: Instrument title: Quality of Life Assessment Visual Analogue scale.Higher scores mean a worse outcome.
  Pain score evaluated POD 1 and POD 2 and Discharge by using a self reported quality of life measure at regular intervals using a visual analog scale (0-10). A higher score means worse outcome and lower score means better outcome.
Time Frame: POD 1 and POD 2 and Discharge
Population: All participants undergoing surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
score on a scale
  POD 1 | 4 [0 to 10] | 4 [0 to 10]
  POD 2 | 3 [0 to 10] | 4 [0 to 10]
  Discharge | 2 [0 to 10] | 3 [0 to 10]

7. Secondary Outcome: Nausea Score
Description: Instrument title: Quality of Life Assessment Visual Analogue scale.Higher scores mean a worse outcome.
  Nausea Score on POD 1 and POD 2 and Discharge by using a self reported quality of life measure at regular intervals using a visual analog scale (0-10). A higher score means worse outcome and lower score means better outcome.
Time Frame: POD 1 and POD 2 and Discharge
Population: All participants undergoing surgery.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
score on a scale
  POD 1 | 1 [0 to 10] | 1 [0 to 10]
  POD 2 | 1 [0 to 10] | 1 [0 to 10]
  Discharge | 1 [0 to 10] | 1 [0 to 10]

8. Secondary Outcome: Bloating Score
Description: Instrument title: Quality of Life Assessment Visual Analogue scale.Higher scores mean a worse outcome.
  Bloating Score on POD 1 and POD 2 and Discharge by using a self reported quality of life measure at regular intervals using a visual analog scale (0-10). A higher score means worse outcome and lower score means better outcome.
Time Frame: POD 1 and POD 2 and Discharge
Population: All participants undergoing surgery.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Clear Liquid Diet | Regular Solid Diet
Number analyzed (Participants) | 50 | 50
score on a scale
  POD 1 | 3 [0 to 10] | 2 [0 to 10]
  POD 2 | 2 [0 to 10] | 2 [0 to 10]
  POD 3 | 2 [0 to 10] | 2 [0 to 10]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Clear Liquid Diet | Regular Solid Diet
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 11/50 | 11/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clear Liquid Diet (N=50) | Regular Solid Diet (N=50)
Post-operative Ileus (Gastrointestinal disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03260426/Prot_SAP_000.pdf